CLINICAL TRIAL: NCT01692236
Title: Neurovascular Magnetic Resonance Imaging in the Assessment of HIV-Associated Neurocognitive Disorders
Brief Title: Brain Imaging for HIV-Associated Thinking and Mood Disorders
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 120200; 12-CC-0200
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2018-04-04

CONDITIONS: Human Immunodeficiency Virus; Neurocognitive Impairment
Keywords: MRI; HIV; Neurocognitive Disorders; Major Depression; Vasculopathy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neurocognitive Disorders; Depressive Disorder, Major; Vascular Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Human immunodeficiency virus (HIV) infection appears to cause problems with blood vessel function. These problems may add to some thinking and mood disorders found in people with HIV infection. Researchers want to evaluate HIV infected patients to see if blood vessel function contributes to thinking and mood disorders, such as early dementia and depression. To do so, they will compare study results between people with and people without HIV infection.

Objectives:

* To compare the thickness of blood vessel walls between people with and without HIV infection.
* To study the relationship between blood vessel thickness and thinking and mood disorders.

Eligibility:

* Individuals between 25 and 55 years of age who have HIV infection.
* Healthy individuals between 25 and 55 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have imaging studies of the brain and major blood vessels in the head and neck.
* Participants will also have neuropsychological testing. These tests will look at memory, learning and thinking ability, attention, and mood.
* Participants will have the option of coming back for repeat blood tests every six months and repeat imaging studies and neuropsychological tests every year, over 1- 4 years period.

DETAILED DESCRIPTION:
With combination antiretroviral therapy, HIV/AIDS has been transformed from a progressive, usually fatal infection to a manageable chronic condition. Yet, HIV associated neurocognitive disorders (HAND) pose a significant clinical problem, even among patients with controlled HIV viremia. There is evidence of accelerated vascular aging and other vascular disorders in HIV-infected (HIV+) people, and studies suggest an association between vascular disorders and unfavorable neurocognitive outcomes. Thus, one possible contributing factor to the high rates of HANDs and depression could be vascular dysfunction, similar to vascular depression and vascular dementia that occur in elderly non-HIV+ individuals. One commonly used diagnostic marker of vasculopathy is thickening of the vessel wall. Multiple studies have already established the correlation between vessel wall thickening and vascular disease manifestations. This prospective observational study aims to examine the relationships between neurocognitive and depression outcomes and vessel wall thickness as a marker of vascular disease in HIV+ adults. We will be using neuropsychological testing, brain imaging, blood biomarkers, and state-of-the-art high-resolution MR imaging of the carotid vessel walls. HIV infected patients (n=40) and HIV-negative controls (n=40) will be recruited. Participants who consent to longitudinal follow-up will be followed for two years with clinical evaluations every 6 months and repeat imaging studies at 12 and 24 months. Cross sectional data analysis will compare markers of vascular and neurocognitive disorders between HIV-infected and HIV-negative participants. The longitudinal data analysis will assess and compare the temporal progression of vascular disease (imaging and blood biomarker findings) in relation to changes in neurocognitive and depression scores in both groups.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for all participants:

1. Age 25-61 years.
2. Willingness to allow stored samples, human leukocyte antigen (HLA) testing, and future genetic testing.
3. Hemoglobin less than or equal to 9.0 g/dL, HCT less than or equal to 28%, platelets less than or equal to 50,000/microL.
4. English language fluency (required for neuropsychological testing).

Additional inclusion criteria for HIV+ participants:

1. Documented HIV infection by standard HIV testing. Prior documentation of HIV- antibody status at the NIH will be accepted in lieu of repeat testing.
2. HIV viral load below the limit of detection on combination antiretroviral therapy for less than or equal to 1 year.
3. Under the care of a primary care physician.

Additional inclusion criteria for HIV-negative participants:

1. HIV-antibody negative.

EXCLUSION CRITERIA:

Exclusion criteria for all participants:

1. Contraindication to MRI scanning, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments.
2. Subjects with a condition precluding entry into scanner and acquisition of scans (e.g., morbid obesity, claustrophobia, back pain, motion disorders).
3. Glomerular filtration rate <45 mL/min/1.73 m(2) as estimated using the Modified Diet in Renal Disease equation.
4. Allergy to qadolinium (MRI contrast)
5. Evidence of current or prior central nervous system opportunistic infection(s) and/or space-occupying lesions such as primary CNS lymphoma.
6. Prior history of intrathecal chemotherapy or radiation therapy to the brain.
7. History of or current diagnosis of systemic vasculitis.
8. Active systemic infection or malignancy requiring therapy.
9. Psychiatric condition interfering with ability to participate in study procedures or provide informed consent.
10. Patient or provider report of alcohol or drug abuse ongoing or within 3 months prior to participation.
11. Sickle cell disease (due to known association with vasculopathy).
12. Systolic blood pressure less than or equal to 180 mmHg at screening.
13. Persons infected with hepatitis C virus (HCV) who are being treated or planning to seek treatment for HCV.
14. Women who are lactating, pregnant, or actively seeking to become pregnant.
15. Other known clinical condition or conditions discovered on MRI that, at the discretion of the investigators, precludes serial clinical, neuropsychological, or imaging evaluation.

Additional exclusion criteria for HIV+ participants

1. HIV acquired perinatally (due to potential effects of HIV and antiretroviral therapy on neurocognitive and vascular development).

Ages: 25 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2012-09-13; Study Completion 2018-04-04

PRIMARY OUTCOMES:
Neuropsychologic testing scores | 1-6 years

SECONDARY OUTCOMES:
Serum biomarkers of cardiovascular disease and inflammation | 1-6 years
MRI brain and vascular findings | 1-6 years

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Connor M. Human immunodeficiency virus (HIV) and stroke: targets for intervention. Infect Disord Drug Targets. 2010 Apr;10(2):76-83. doi: 10.2174/187152610790963483. PMID 20166974
- [Background] Highleyman L. Mortality trends: toward a new definition of AIDS? BETA. 2005 Winter;17(2):18-28. PMID 15828120
- [Background] Holtgrave DR. Causes of the decline in AIDS deaths, United States, 1995-2002: prevention, treatment or both? Int J STD AIDS. 2005 Dec;16(12):777-81. doi: 10.1258/095646205774988109. PMID 16336756